CLINICAL TRIAL: NCT05992870
Title: Neoadjuvant Radiotherapy and Immediate Implant-Based Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xinhong Wu, PhD, vice-president, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoRTIBR
Record Dates: First submitted 2023-08-05; First posted 2023-08-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Implant Breast Reconstruction; Neoadjuvant Radiotherapy
Keywords: neoadjuvant radiotherapy, implant, breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant radiotherapy group (Experimental): Radiotherapy followed by skin-sparing mastectomy and immediate implant-based reconstruction in HBCH
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — In case of neoadjuvant chemotherapy, RT will start 3-4 weeks after the last course of chemotherapy. A dose of 15 x 2.67 Gy 5 fractions or 16 x 2.67Gy 5 fractions per week.
  A skin-sparing mastectomy and a immediate implant-based breast reconstruction will be performed, approximately 2-6 weeks after latest radiotherapy treatment.

SUMMARY:
Neoadjuvant radiotherapy(NART) followed by mastectomy and immediate DIEP flap reconstruction is feasible and technically safe. However, reports of NACT followed immediate implant-based breast reconstruction are rare. Some studies have shown that NART followed immediate implant-based breast reconstruction seems feasible and can be safely attempted. It's well known that radiotherapy after implant-based breast reconstruction have negative effects on implant and cosmetic results. So, investigators conducted a polit study to learn about acute post-surgical complications following skin-sparing mastectomy and immediate implant-based breast reconstruction after NART.

DETAILED DESCRIPTION:
Radiotherapy after implant-based breast reconstruction have negative effects on implant and cosmetic results, including severe capsular contracture, mastectomy flap necrosis ,reoperation and so on. Postmastectomy radiotherapy( PMRT )is associated with implant reconstruction failure. PRADA study has shown neoadjuvant radiotherapy followed by skin-sparing mastectomy and immediate DIEP flap reconstruction is feasible and technically safe. The investigators assume that neoadjuvant radiotherapy can avoid the negative effects of PMRT on an implant and the capsule of an implant and would lead to better cosmetic results and less complications compared to PMRT. Furthermore, some studies have shown that NART could potentially result in shorter time between diagnosis and treatment completion. So, investigators conducted a polit study to learn about acute post-surgical complications following skin-sparing mastectomy and immediate implant-based breast reconstruction after NART.

ELIGIBILITY:
Inclusion Criteria:

Women >18 years with histopathologically-confirmed breast cancer, who:

* require mastectomy for any reason
* a known indication for (adjuvant) radiotherapy
* require implant-based breast reconstruction

Exclusion Criteria:

* Inability to give informed consent
* MDT unable to make recommendation for radiotherapy based on pre-operative histopathological and imaging findings
* Previous history of breast cancer or another malignancy for which radiotherapy of the breast or axilla
* Pregnant or lactating
* inflammatory breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-08 (Actual); Primary Completion 2025-07-08 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications at 3 months following skin-sparing mastectomy and immediate implant-based breast reconstruction after NART | 3 months following skin-sparing mastectomy and immediate breast reconstruction
  Surgical complications are defined as any complication requiring surgical intervention necessary within a period up to three months after the final reconstruction. Including Infection, hematoma , loss of implant or flap, fat necrosis, wound breakdown,defined and scored using the C-DC37.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 . | Within 3 months after both breast reconstruction and radiotherapy
  Other adverse events following NART or surgery other than described in the primary outcome measure.
Number of participants with removal of implant. | 6 months after surgery
  Implant are removed for postoperative complications.
Patient satisfaction. | 3 months and 12 months after surgery
  Patient satisfaction (as measured using the BREAST-Q reconstruction module) before, 3 months after, and 12 months after surgery.
Pathological complete response (pCR) assessed in skin-sparing mastectomy specimen | Within 2 weeks after skin-sparing mastectomy
  A pCR was defined as absence of invasive and in situ carcinoma in the breast, irrespective of nodal status (ypT0).

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhong Wu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF)